CLINICAL TRIAL: NCT01903720
Title: A Safety and Efficacy Study of OZURDEX® in Macular Edema Associated With Branch Retinal Vein Occlusion
Acronym: COBALT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APMA-OZU-01-01
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OZURDEX® (Experimental): OZURDEX® (700 µg dexamethasone implant) administered intravitreally on day 0, and approximately every 4 months as needed (based on physician judgment) for up to 12 months.
  Interventions: Drug: dexamethasone implant

INTERVENTIONS:
Drug: dexamethasone implant — OZURDEX® (700 µg dexamethasone implant) administered intravitreally on day 0, and approximately every 4 months as needed (based on physician judgment) for up to 12 months.
  Other Names: OZURDEX®

SUMMARY:
This study will evaluate the safety and efficacy of OZURDEX® (700 µg dexamethasone implant) in patients with macular edema associated with branch retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of macular edema
* Best corrected visual acuity of approximately 20/400 to 20/40 in the study eye

Exclusion Criteria:

* Use of systemic steroids (eg, oral, intravenous, intramuscular, epidural, rectal, or extensive dermal) within 1 month
* Intraocular surgery, including cataract surgery, and/or laser surgery of any type within 3 months
* Any active ocular infection in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-07-16 (Actual); Primary Completion 2014-09-24 (Actual); Study Completion 2015-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Seoul, South Korea

REFERENCES:
- [Background] Yoon YH, Kim JW, Lee JY, Kim IT, Kang SW, Yu HG, Koh HJ, Kim SS, Chang DJ, Simonyi S. Dexamethasone Intravitreal Implant for Early Treatment and Retreatment of Macular Edema Related to Branch Retinal Vein Occlusion: The Multicenter COBALT Study. Ophthalmologica. 2018;240(2):81-89. doi: 10.1159/000487547. Epub 2018 Apr 11. PMID 29642062

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OZURDEX®
Started | 71
Completed | 59
Not Completed | 12
Not completed — Inclusion / exclusion criteria not met | 6
Not completed — Adverse Event | 1
Not completed — Rescinding of informed consent | 2
Not completed — Lost to Follow-up | 2
Not completed — Treatment with alternative drug | 1

BASELINE CHARACTERISTICS:
Arm/Group | OZURDEX®
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.46 (9.19)
Age, Customized [Number; unit: participants]
  30 to 39 years | 1
  40 to 49 years | 12
  50 to 59 years | 29
  60 to 69 years | 22
  70 years and over | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) at Month 6
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly ranging from 0 (worst) to 100 letters (best). A positive number change in the number of letters read correctly means that the vision improved and a negative number change in the number of letters read correctly means that the vision has worsened.
Time Frame: Baseline, Month 6
Population: Intent-to-treat (ITT) population included all enrolled participants. "n" in the category is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | OZURDEX®
Number analyzed (Participants) | 71
letters
  Baseline | 51.90 (13.55)
  Change from Baseline at Month 6 (n=62) | 18.60 (12.90)

2. Secondary Outcome: Change From Baseline in Central Retinal Thickness (CRT) at Month 6
Description: CRT was measured in the study eye using optical computed tomography (OCT), a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina. A negative change from Baseline indicates an improvement.
Time Frame: Baseline, Month 6
Population: ITT population included all enrolled participants. "n" in the category is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Arm/Group | OZURDEX®
Number analyzed (Participants) | 71
micrometers (μm)
  Baseline | 505.13 (129.91)
  Change from Baseline at Month 6 (n=62) | -246.82 (150.74)

3. Secondary Outcome: Change From Baseline in BCVA at Month 12
Description: as for outcome 1
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | OZURDEX®
Number analyzed (Participants) | 71
letters
  Baseline | 51.90 (13.55)
  Change from Baseline at Month 12 (n=59) | 15.27 (14.99)

4. Secondary Outcome: Change From Baseline in CRT at Month 12
Description: as for outcome 2
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | OZURDEX®
Number analyzed (Participants) | 71
μm
  Baseline | 505.13 (129.91)
  Change from Baseline at Month 12 (n=59) | -196.90 (164.07)

5. Secondary Outcome: Change From Baseline in BCVA at Each Visit
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly ranging from 0 (worst) to 100 letters (best). A positive number change in the number of letters read means that the vision improved and a negative number change in the number of letters read means that the vision has worsened.
Time Frame: Baseline, Week 1, Months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
Population: ITT population included all enrolled participants. "n" in the category is the number of participants with data available at the given time-point for analysis.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | OZURDEX®
Number analyzed (Participants) | 71
letters
  Baseline | 51.90 (13.55)
  Change from Baseline at Week 1 (n=70) | 12.80 (10.69)
  Change from Baseline at Month 1 (n=66) | 16.08 (10.75)
  Change from Baseline at Month 2 (n=62) | 18.84 (12.16)
  Change from Baseline at Month 3 (n=63) | 17.59 (12.90)
  Change from Baseline at Month 4 (n=59) | 14.37 (13.47)
  Change from Baseline at Month 5 (n=63) | 18.10 (13.44)
  Change from Baseline at Month 6 (n=62) | 18.60 (12.90)
  Change from Baseline at Month 7 (n=60) | 18.02 (12.64)
  Change from Baseline at Month 8 (n=61) | 16.02 (13.39)
  Change from Baseline at Month 9 (n=59) | 15.88 (13.35)
  Change from Baseline at Month 10 (n=60) | 17.68 (13.17)
  Change from Baseline at Month 11 (n=59) | 15.54 (14.04)
  Change from Baseline at Month 12 (n=59) | 15.27 (14.99)

6. Secondary Outcome: Change From Baseline in CRT at Each Visit
Description: as for outcome 2
Time Frame: Baseline, Week 1, Months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Arm/Group | OZURDEX®
Number analyzed (Participants) | 71
micrometers (μm)
  Baseline | 505.13 (129.91)
  Change from Baseline at Week 1 (n=70) | -173.67 (140.57)
  Change from Baseline at Month 1 (n=66) | -229.48 (142.45)
  Change from Baseline at Month 2 (n=62) | -255.55 (139.01)
  Change from Baseline at Month 3 (n=63) | -188.17 (179.84)
  Change from Baseline at Month 4 (n=59) | -100.76 (150.97)
  Change from Baseline at Month 5 (n=63) | -202.41 (157.66)
  Change from Baseline at Month 6 (n=62) | -246.82 (150.74)
  Change from Baseline at Month 7 (n=60) | -220.13 (143.07)
  Change from Baseline at Month 8 (n=60) | -175.83 (133.93)
  Change from Baseline at Month 9 (n=59) | -211.46 (158.10)
  Change from Baseline at Month 10 (n=59) | -250.97 (133.24)
  Change from Baseline at Month 11 (n=59) | -219.14 (144.47)
  Change from Baseline at Month 12 (n=59) | -196.90 (164.07)

7. Secondary Outcome: Percentage of Participants With a Change From Baseline of 15 or More Letters in BCVA
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly ranging from 0 (worst) to 100 letters (best). An increase in the number of letters read correctly means that the vision improved and a decrease in the number of letters read correctly means that the vision has worsened.
Time Frame: Baseline, Months 6 and 12
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | OZURDEX®
Number analyzed (Participants) | 62
percentage of participants
  Month 6_Increase | 64.52
  Month 6_Decrease | 1.61
  Month 12_Increase (n=59) | 55.93
  Month 12_Decrease (n=59) | 5.08

8. Secondary Outcome: Percentage of Participants Receiving a Second Injection
Time Frame: 12 Months
Population: ITT population included all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | OZURDEX®
Number analyzed (Participants) | 71
percentage of participants | 18.31

9. Secondary Outcome: Percentage of Participants Receiving a Third Injection
Time Frame: 12 Months
Population: ITT population included all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | OZURDEX®
Number analyzed (Participants) | 71
percentage of participants | 49.30

10. Secondary Outcome: Time to Second Injection
Description: Time in weeks from the first injection to the second injection.
Time Frame: 12 Months
Population: ITT population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | OZURDEX®
Number analyzed (Participants) | 71
weeks | 20.78 (6.02)

11. Secondary Outcome: Time to Third Injection
Description: Time in weeks from the second injection to the third injection.
Time Frame: 12 Months
Population: ITT population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | OZURDEX®
Number analyzed (Participants) | 71
weeks | 19.20 (3.09)

12. Secondary Outcome: Percentage of Participants Who Received Laser Treatments
Description: Participants underwent laser photocoagulation therapy for all areas of foveal leakage and non-perfusion, as well as areas of extensive retinal hyperplasia if applicable for rescue therapy.
Time Frame: 12 Months
Population: ITT population included all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | OZURDEX®
Number analyzed (Participants) | 71
percentage of participants | 0.0

ADVERSE EVENTS:
Arm/Group | OZURDEX®
Serious Adverse Events (participants affected / at risk) | 2/71
Other Adverse Events (participants affected / at risk) | 44/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OZURDEX® (N=71)
Cataract (Eye disorders) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OZURDEX® (N=71)
Dry eye (Eye disorders) | 14
Cataract (Eye disorders) | 12
Conjunctival haemorrhage (Eye disorders) | 8
Vitreous detachment (Eye disorders) | 4
Intraocular pressure increased (Investigations) | 25
Headache (Nervous system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.